CLINICAL TRIAL: NCT04837469
Title: Randomized Clinical Trial of Fissure Sealants Comparing Universal Adhesive With Etch-And-Rinse Adhesive After 24 Month
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Dr Emel Karaman, associate professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2014/743
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Fissure, Dental; Adhesion
Keywords: fissure sealant, adhesive
MeSH Terms: conditions — Dental Fissures; Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Universal Adhesive (Experimental): universal adhesive
  Interventions: Procedure: fissure sealant application
- Etch-And-Rinse Adhesive (Experimental): Etch-And-Rinse Adhesive
  Interventions: Procedure: fissure sealant application

INTERVENTIONS:
Procedure: fissure sealant application — fissure sealants were placed after differnt adhesive strategies used

SUMMARY:
Objective: This randomized, controlled clinical study aimed to evaluate the performance of one universal adhesive applied with etch-and-rinse or self-etch strategy and one etch-and-rinse adhesive on fissure sealant retention over 24 months. Methodology: 144 sealants were placed on the permanent premolars and molars of 13 subjects. Teeth were divided into three groups SB2(control): Adper Single Bond 2, SBU-ER: Single Bond Universal/etch-and-rinse, SBU-SE: Single Bond Universal/self-etch. After the adhesive application, Fissurit FX was applied and light-cured. Clinical evaluations were done at baseline and at 1 week, 6-, 12-, 18- and 24-month recalls. Visual examination was performed on every visit for evaluation of the sealants. Evaluating criteria were: 1= completely retained; 2= partial loss; 3= total loss. The Pearson Chi-square test was used for each evaluation period.

DETAILED DESCRIPTION:
Thirteen patients with a mean age of 20.5 (range 19-22) were selected among the patients seeking routine dental care from Conservative Dentistry Department who met the inclusion criteria. Inclusion criteria were: good oral hygiene and and the absence of caries, previously placed restorations, bruxism and an allergy to the materials tested.

Bitewing radiographs were taken. Pellicle and any remaining plaque on the fissures were removed by using slurry of pumice with a slow-speed handpiece. All restorative procedures were performed by the same operator. The teeth were assigned for different group by using a table of random numbers.

Group 1 (SB2): Etched with 35% phosphoric acid gel for 30 s, rinsed and dried. Adper Single Bond 2 (3M ESPE St. Paul MN. USA) applied and light cured for 10s with a LED device (Demi Plus; Kerr, Switzerland) Group 2 (SBU-ER) : Etched with 35% phosphoric acid gel for 30s, rinsed and dried. Single Bond Universal Adhesive (3M ESPE St. Paul MN.USA) applied, gently air thinned for 5 s and light cured for 10s with a LED device Group 3 (SBU-SE): Single Bond Universal Adhesive (3M ESPE St. Paul MN.USA) applied for 20 s with vigorous agitation, gently air thinned for 5 s and light cured for 10 s with a LED device A nanofilled fissure sealant, Fissurit FX (Voco,Cuxhaven,Germany) was applied to the fissures and air entrapment was prevented by carefull spreading with a dental probe. The sealant material was light-cured for 20 seconds with LED. The occlusion was checked with articulating paper. Fine-grit diamond burs (Diatech, Swiss Dental, Switzerland) and rubber cups (Edenta AG, AU SG, Switzerland). were used for finishing and polishing.

Each restoration was evaluated at baseline,1week after treatment and 6, 12, 18 and 24 months. Evaluation of restorations was carried out by two calibrated examiners who were unaware of group allocation and who were not involved with the treatment procedures, by the help of a mirror, blunt explorer and air stream. Caries formation was evaluated as present or absent and the sealants were evaluated according to the following criteria: 1= Completely retained 2= Partial loss 3= Total loss.

ELIGIBILITY:
Inclusion Criteria:

* good oral hygiene and and the absence of caries, previously placed restorations, bruxism and an allergy to the materials tested.

Exclusion Criteria:

* bad oral health, maloclusion, allergy to resins used

Ages: 19 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-02-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
The evaluation of retention rate of fissure sealants | 24 month

IPD SHARING:
Plan to Share IPD: No